CLINICAL TRIAL: NCT04378621
Title: Treatment of Inflammation Versus Hand Training to Prevent and Revert Neuropsychiatric Comorbidity in Patients With Rheumatoid Arthritis
Brief Title: Effect of Antiinflammatory Treatment Versus Hand Training on Neuropsychiatric Comorbidity in RA-patients
Acronym: NeuMRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuMRA
Record Dates: First submitted 2020-04-08; First posted 2020-05-07 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Pain; Fatigue; Cognitive Decline; Depression; Brain Diseases; Hand Rheumatism
Keywords: Rheumatoid arthritis; RA; neuropsychiatric comorbidity
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain; Fatigue; Cognitive Dysfunction; Depression; Brain Diseases | interventions — Janus Kinase Inhibitors; Etanercept; Infliximab; Adalimumab; Certolizumab Pegol; golimumab; baricitinib; tofacitinib

STUDY DESIGN:
Intervention Model Description: Group A. Pharmacological treatment with TNF-α inhibitor or JAK inhibitor Group B. Physical hand training 10 min twice daily while on stable treatment with TNF-α inhibitor or JAK inhibitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacological anti-inflammatory treatment (Experimental): Use of anti-rheumatic treatment with TNF-α inhibitor (subcutaneous injection given once or twice a week) or JAK inhibitor (per oral tablet once or twice a day)
  Interventions: Drug: TNF-α inhibitor OR JAK inhibitor
- Physical hand training (Experimental): Physical hand training 10 min twice daily while on stable treatment
  Interventions: Other: Hand training

INTERVENTIONS:
Drug: TNF-α inhibitor OR JAK inhibitor — Pharmacological anti-rheumatic treatment
  Other Names: TNF-a inhibitors: Etanercept (Enbrel, Benapali), Infliximab (Remicade, Inflectra, Flixabi), Adalimumab (Humira, Imraldi, AMGEVITA), Certolizumabpegol (Cimzia), Golimumab (Simponi); JAK-inhibitors: Baricitinib (Olumiant), Tofacitinib (Xeljanz)
  Arms: Pharmacological anti-inflammatory treatment
Other: Hand training — Physical hand training 10 min twice daily while on stable treatment
  Other Names: physiotherapy of hands
  Arms: Physical hand training

SUMMARY:
The purpose of this study is to investigate how RA affect the brain structures in RA-patients and if anti-inflammatory treatment that target TNF-α or JAK OR physical training of hands has positive impact on neuropsychiatric symptoms and morphological changes in the brain caused by the disease.

The goal of this research project is to improve the knowledge of morphological changes in brain developed in connection to RA and to identify clinical and serological markers to predict development of those changes and finally, to investigate if anti-rheumatic interventions counteract destructive processes in the central nervous system (CNS) and improve the patient's health with respect to functionality, pain experience and psychological well-being.

DETAILED DESCRIPTION:
Based on the information gained in previous studies the investigators want to examine if;

A. anti-inflammatory treatment that target TNF-α or JAK signalling or

B. physical training of hands

has a positive impact on neuropsychiatric symptoms and morphological changes in the brain caused by RA.

To examine this the investigators will employ a prospective open-label study design with two parts, one observation part (1) and one intervention part (2). Patients will be assigned to either:

1. OBSERVATION PART

Aim: Mapping brain morphology in relation to functional impairment, inflammation and neuropsychiatric symptoms in patients with RA of various disease duration.

To study this 80 RA patients will be recruited from the outpatient clinic at Sahlgrenska university hospital for an observational prospective study.

RA-patients will be identified via the diagnosis registry within Reumatologi/Sahlgrenska Universitetssjukhuset.

Inclusion criteria: patients age 45-75 years; confirmed RA diagnosis, in the early stage of the disease (1-3 years after the diagnosis, n=20); in the established stage of the disease (5-8 years after the diagnosis, n=30) and in the late stage of the disease (>12 years after the diagnosis, n=30).

Exclusion criteria: any conditions precluding MRI imaging; e.g claustrophobia; pacemaker etc, medical history of ischemic stroke or cerebral hemorrhage; medical history of neurological disease; inability to read and communicate in Swedish, hence being able to give informed consent and fill out study questionnaires.

The patient will then undergo the study related activities; clinical examination by rheumatologist and occupational therapist, blood sampling, height and weight, waist circumference, blood pressure measurement, questionnaires (see below and attachment), plain radiological imaging of hands and MRI of the head.

1. * Clinical examination:

   * Documentation of number of tender and swollen joints according to the established Disease Activity Score 28-protocol (DAS28) (see attachment DAS28).
   * Documentation of number of Tender Points ie sensitive areas on the body that become painful when pressure is applied according to the established TP 18 protocol (see attachment TP18).
   * Documentation of the hand joint mobility,
   * pain (VAS), grip strength,
   * Functional arm-shoulder-hand status according to DASH protocol (see attachment Handstatus).
   * Questionnaires used in the study are:

   the Health Assessment Questionarie (HAQ), the Fibromyalgia Questionaire (FIQ), the Hospital Anxiety and Depression Scale (HADS) (HADS), the Short Form Health Survey (SF-36), the IPAQ (International Physical Activity Questionnaire), the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. Questions on the patients´ diagnosis and pharmacological treatment (and for women questions on hormonal status) and tobacco habits are also collected.
   * Radiological imaging of hands
   * Anatomical 3D MRI of the head will be performed using a standard protocol of T1-weighted 3D scan with approximately isotropic voxels and a resolution of approximately 1 mm^3 per voxel. The field of view (FOV) will include the head in full and extend caudally to include the cerebellum and medulla. Automatic anatomical segmentation using MAPER (multi-atlas propagation with enhanced registration) will be applied.
2. INTERVENTION PART

Aim: To study the effect of TNF-α inhibitors/JAK inhibitors and regular physical training of hands on RA-related intracranial changes. Based on the information gained in the cross-sectional and in the pilot part of the investigators previous studies (Erlandsson 2016; Andersson 2018), they want to investigate if anti-inflammatory treatment that target TNF-α or JAK OR physical training of hands has a positive impact on neuropsychiatric symptoms and morphological changes in the brain caused by RA.

To examine this a prospective open-labeled study with two groups with 66 patients in each group will be employed.

Patients will be assigned to either:

Group A. Pharmacological treatment with TNF-α inhibitor or JAK inhibitor

Group B. Physical hand training 10 min twice daily while on stable treatment with TNF-α inhibitor or JAK inhibitor

Inclusion criteria: patients age 45-75 years; confirmed and established RA. Naïve to treatment with TNF-α inhibitors or JAK inhibitors to be eligible for Group A and to be on a stable treatment of TNF-α inhibitors or JAK inhibitors for the last 3 months to be eligible for Group B.

Exclusion criteria: other serious conditions precluding MRI imaging, claustrophobia; medical history of ischemic stroke or cerebral hemorrhage; medical history of neurological disease; inability to read and communicate in Swedish, hence being able to give informed consent and fill out study questionnaires.

For Group A, RA patients attending the outpatient clinic at Sahlgrenska university hospital set to start treatment with TNF-α inhibitors or JAK inhibitors for the first time will be included. Both TNF-α inhibitors and JAK inhibitors are well tolerated, efficient anti-rheumatic drugs administered to RA patients with moderate to severe disease in accordance with the current recommendations for pharmacological treatment of RA (www.svenskreumatologi.se/srfs-riktlinjer/#).

For Group B, RA patients who already receive stable treatment with TNF-α or JAK inhibitors since 3 months will be included. These patients will be instructed to carry out hand exercises designed by an occupational therapist for 10 min twice daily for the entire study period of 6 months (training program attached).

Patients fulfilling the inclusion criteria are informed of the study by their responsible rheumatologist. Before approaching the patient, the doctor will have made sure he/she fulfils the study criteria and that he/she is susceptible and open for information about a clinical study. The decision to start treatment with TNF-α or JAK inhibitors will be made by a rheumatologist on the intention to treat basis, completely outside the scope of this study. We will not in any way affect this decision, but simply recruit patients from those that are starting TNF-α or JAK inhibitors. Once the patient has received information about the study, both orally and in text, and has been given time to think and ask questions, they are asked to participate and if so sign the informed consent. After consent is signed by both patient and personnel a copy is given to the patient.

The patient will then undergo the study related activities; clinical examination by rheumatologist and occupational therapist, blood sampling, height, weight, waist circumference and blood pressure measurement, completion of study questionnaires (see below and attachment), plain radiological imaging of hands and MRI of the head. Information regarding RA duration, clinical activity and medication will be retrieved from medical records.

1. Clinical examination:

   * Documentation of number of tender and swollen joints according to the established Disease Activity Score 28-protocol (DAS28) (see attachment DAS28).
   * Documentation of number of Tender Points, ie sensitive areas on the body that become painful when pressure is applied according to the established TP 18 protocol (see attachment TP18).
   * Documentation of the hand joint mobility,
   * pain (VAS),
   * Grip strength,
   * Functional status in shoulder, arm and hand according to DASH (see attachment Handstatus).
2. Anatomical 3D MRI of the head will be performed using a standard protocol of T1-weighted 3D scan with approximately isotropic voxels and a resolution of approximately 1 mm^3 per voxel. The field of view (FOV) will include the head in full and extend caudally to include the cerebellum and medulla.
3. Radiological imaging of hands
4. The study participants of both groups will write a pain diary to register pain (by visual analogue scale) on daily basis (attached).

For all patients participating in the interventional part of study, both group A and B, follow-up visits 3 and 6 months after first visit will be booked. At these visit they will meet with occupational therapist for assessment of hand function, leave blood, complete study questionnaires and hand over their completed pain diary. At the 6 month-visit an anatomic 3D MRI of the head will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* confirmed RA diagnosis, in the early stage of the disease (1-3 years after the diagnosis, n=20); in the established stage of the disease (5-8 years after the diagnosis, n=30) and in the late stage of the disease (>12 years after the diagnosis, n=30)

Exclusion Criteria:

* any conditions precluding MRI imaging; e.g claustrophobia; pacemaker etc, medical history of ischemic stroke or cerebral hemorrhage; medical history of neurological disease; inability to read and communicate in Swedish, hence being able to give informed consent and fill out study questionnaires

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in regional brain volume | Difference in brain regional volume from base-line to follow-up study visit after 6 months
  Magnetic resonance imaging (MRI) of all patients brains will be performed at base-line and at follow-up visit after 6 months. Measurement of 83 anatomical regions of the brain will be performed to detect subtle changes in volume. This is performed using multiatlas propagation with enhanced registration (MAPER) and the 2017 version of the Hammersmith atlas database.
  The difference in regional brain volume between study visits will be calculated.
Difference in Disease activity score (DAS28) | Difference in DAS28 score from base-line to follow-up study visit after 6 months
  Scoring of disease activity for all patients will be performed at base-line and at follow-up visit after 6 months. Disease Activity Score is a standardised indicator of RA disease activity calculated as a composite score of: number of tender and swollen joints (assessed by trained personnel), erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) and the patients assessment of pain on a visual analogue scale of 10 mm (VAS).
  The difference in Disease activity score between study visits will be calculated.
Difference in Tender Point score (TP18) | Difference in TP18 score from base-line to follow-up study visit after 6 months
  Scoring of tender Points for all patients will be performed at base-line and at follow-up visit after 6 months. Tender points are sensitive areas on the body that elicit pain and tenderness when pressure is applied. The TP 18 protocol is a standardised measurement of number of painful/tender points out of 18 bilateral points on the body.
  The difference in Tender Point score between study visits will be calculated.
Difference in Pain VAS score | Difference in Pain VAS score from base-line to follow-up study visit after 3 and 6 months
  Scoring of Pain VAS will be performed daily by all patients and recorded in a pain diary. Pain VAS is the patients scoring in mm of overall perceived pain on a 10 mm long visual analogue scale.
  The difference in Pain VAS score between daily recordings will be calculated.
Difference in hand joint mobility | Difference in hand joint mobility from base-line to follow-up study visits after 3 and 6 months
  Measurement of hand joint mobility for all patients will be performed at base-line and at follow-up visit after 3 and 6 months. Hand joint mobility is clinically assessed by occupational therapist according to a standardised protocol and reported as degrees of mobility in extension/flexion and pronation/supination of the hand joint.
  The difference in degrees of hand joint mobility between study visits will be calculated.
Difference in finger joint mobility | Difference in finger joint mobility from base-line to follow-up study visits after 3 and 6 months
  Measurement of finger joint mobility for all patients will be performed at base-line and at follow-up visit after 3 and 6 months. Finger joint mobility is clinically assessed by occupational therapist according to standardised protocol and reported as degrees of mobility in extension/flexion of each finger.
  The difference in degrees of finger joint mobility between study visits will be calculated.
Difference in hand grip strength | Difference in hand grip strength from base-line to follow-up study visits after 3 and 6 months
  Measurement of hand grip strength for all patients will be performed at base-line and at follow-up visit after 3 and 6 months. Hand grip strength is clinically assessed by occupational therapist and performed using Grippit®, a standardised electronic handheld instrument used for measuring hand strength in the cylinder grip.
  The patient is instructed to grip the Grippit® and squeeze it as hard as possible for 10 seconds. The instrument generates three values; the maximal value of force applied, the mean value of force applied during the 10 seconds and a final value measured during the last half a second. The values are reported in Newton (N). Both hands are examined and which of the hands that is dominant is noted.
  The difference in Newton between study visits will be calculated.
Difference in hand/finger joint deformities | Difference in hand/finger joint deformities from base-line to follow-up study visits after 3 and 6 months
  Documentation of hand/finger joint deformities for all patients will be performed at base-line and at follow-up visit after 3 and 6 months. Hand and finger joint deformities is clinically assessed by occupational therapist according to standardised protocol.
  Reported in text for each joint
Difference in RA-related skeletal changes | Difference in RA-related skeletal changes from base-line to follow-up study visits after 6 months
  Documentation of RA-related skeletal changes for all patients will be performed at base-line and at follow-up visit after 6 months. Radiological imaging of the hand joint will be performed using plain X-ray. The assessment of hand radiographs and scoring of possible joint damage will be performed by experienced rheumatologist.
  The difference in score between study visits will be calculated.
Difference in inflammatory markers | Difference in inflammatory markers from base-line to follow-up study visits after 3 and 6 months
  Serum samples will be gathered from all patients at base-line and follow-up visit after 3 and 6 months. Levels of various inflammatory markers will be measured and the difference in levels between study visits will be calculated.
Difference in DASH score | Difference in DASH score from base-line to follow-up study visits after 3 and 6 months
  DASH, "Disabilities of the Arm, Shoulder and Hand", is a self-administered questionnaire regarding symptoms and ability to perform certain activities. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in DASH score between study visits will be calculated.
Difference in FIQ score | Difference in FIQ score from base-line to follow-up study visits after 3 and 6 months
  FIQ, "Fibromyalgia Impact Questionnaire", is a self-administered questionnaire regarding pain, fatigue, functional ability, quality of life etc. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in FIQ score between study visits will be calculated.
Difference in HADS score | Difference in HADS score from base-line to follow-up study visits after 3 and 6 months
  HADS, "Hospital Anxiety and Depression Scale", is a self-administered questionnaire regarding anxiety and depression. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in HADS score between study visits will be calculated.
Difference in IPAQ score | Difference in IPAQ score from base-line to follow-up study visits after 3 and 6 months
  IPAQ, "International Physical Activity Questionnaire", is a self-administered questionnaire regarding physical activity and inactivity. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in IPAQ score between study visits will be calculated.
Difference in HAQ score | Difference in HAQ score from base-line to follow-up study visits after 3 and 6 months
  HAQ, "Health Assessment Questionnaire", is a self-administered questionnaire regarding functional ability and overall health. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in HAQ score between study visits will be calculated.
Difference in SF-36 score | Difference in SF-36 score from base-line to follow-up study visits after 3 and 6 months
  SF-36, "Short Form Health Survey", is a self-administered questionnaire regarding overall health. The questionnaire will be filled out by all patients at base-line and at follow-up visit after 3 and 6 months and scored according to established protocol.
  The difference in SF-36 score between study visits will be calculated.

SECONDARY OUTCOMES:
Difference in intestinal microbiome composition | Difference in intestinal microbiome composition from base-line to follow-up study visits after 6 months
  Fecal sample will be gathered from all patients at base-line and follow-up visit after 6 months.
  Analyses of the microbiome composition will be performed and difference in data between study visits will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bokarewa, MD, Principal Investigator — Dep of Rheumatology and Inflammation research, University of Gothenburg, Sweden
Locations (1):
- Clinical Rheumatology Research Center (CRRC), Department of Rheumatology, Sahlgrenska University Hospital, Gothenburg, Sweden